CLINICAL TRIAL: NCT03907787
Title: The Use of a New Food-grade Lecithin Formulation of Highly Standardized Ginger (Zingiber Officinale) and Acmella Oleracea Extracts for the Treatment of Pain and Inflammation in a Group of Subjects With Moderate Knee Osteoarthritis
Brief Title: Zingiber and Acmella Against Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206/15012017
Record Dates: First submitted 2019-03-26; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Pain; Osteo Arthritis Knee
MeSH Terms: conditions — Pain | interventions — ginger extract

STUDY DESIGN:
Intervention Model Description: One-group pretest-posttest quasi-experimental design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One-group pretest-posttest quasi-experimental design (Other): 50 subjects with moderate knee osteoarthritis were supplied for four weeks with two tablets/day, each containing 350 mg of standardized extracts of Zingiber officinale and Acmella oleracea.
  Interventions: Dietary Supplement: Zingiber officinale and Acmella oleracea

INTERVENTIONS:
Dietary Supplement: Zingiber officinale and Acmella oleracea — Subjects were supplied for four weeks with two tablets/day and there was the evaluation of pain intensity, by a 30-days Visual Analogue Scale (VAS) and b) the assessment of knee function by Western Ontario and McMaster Universities Arthritis Index and by Tegner Lysholm Knee Scoring collected at baseline, at 15 and 30 days after treatment, Health-related quality of life, by the ShortForm36, inflammation by C-reactive protein and Erythrocyte Sedimentation Rate, body composition by dual-energy X-ray absorptiometry measured at baseline and 30 days after treatment.

SUMMARY:
One-group pretest-posttest quasi-experimental design in which primary outcomes were: a) the evaluation of pain intensity, by a 30-days Visual Analogue Scale (VAS) and b) the assessment of knee function by Western Ontario and McMaster Universities Arthritis Index and by Tegner Lysholm Knee Scoring collected at baseline, at 15 and 30 days after treatment. Secondary outcomes were the evaluation: c) of Health-related quality of life, by the ShortForm36, d) of inflammation by C-reactive protein and Erythrocyte Sedimentation Rate, and e) of body composition by dual-energy X-ray absorptiometry measured at baseline and 30 days after treatment.

DETAILED DESCRIPTION:
To evaluate the safety and the efficacy on pain and inflammation of a new food-grade lecithin formulation of standardized extracts of Zingiber officinale and Acmella oleracea.

ELIGIBILITY:
Inclusion Criteria:

* established moderate knee OA (classification 1-3 according to Kellgren and Lawrence system for classification of knee OA)
* Lequesne Index of 6-10; 3) Body Mass Index (BMI) between 22 and 30 kg/m2
* aged 40-75
* no drugs for OA, such as nonsteroidal anti-inflammatory drugs (NSAIDs).

Exclusion Criteria:

* diabetes, metabolic disease, or neoplasia, as well as the patients with disabling diseases that could directly affect muscle weakness (such as neurological diseases, hip fractures, or amputations)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Change in generic pain (Visual Analogue Scale) | 0-15-30 days
  Pain intensity measured both at motion and at rest, using the Visual Analogue Scale (VAS). VAS measures a characteristic or attitude ranging across a continuum of values and cannot be directly measured. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks. The results are showed with a scale 0-10. 0 means no pain and 10 high pain.
Change in knee pain (WOMAC) | 0-15-30 days
  Assessment of knee pain by WOMAC (Western Ontario and McMaster Universities Arthritis) Index. The WOMAC pain scale consists of five questions that assess pain while walking on a flat surface, going up or down stairs, in bed at night, sitting or lying, and standing upright. The responses are recorded on a five-point Likert scale, with a higher score representing a greater level of pain. This scale is valid and reliable in hip and knee OA populations.
Change in knee functionality (TLKS) | 0-15-30 days
  Tegner Lysholm Knee function Scoring (TLKS). Each patient completed a self-report questionnaire, TLKS, related to knee symptoms and function. It includes eight items: Limp, Support, Locking, Instability, Pain, Swelling, Stair climbing and Squatting. Each possible response to the items gives an arbitrary score on an increasing scale with a maximum of 100, a higher score representing a higher ability.

SECONDARY OUTCOMES:
Change Health-related quality of life: ShortForm36 | 0-30 days
  Health-related quality of life, recorded by the Short Form 36 Health questionnaire (SF-36), a generic measure of health status designed for use in population surveys which consider body pain as a dimension of health status. This is a self-reporting questionnaire and outcomes are measured with 8 numbers that express 8 different aspects of quality of life. Scoring 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the given scoring key. all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered.
Change in inflammatory blood markers (CRP) (mg/dl) | 0-30 days
  Inflammation markers in plasma: C-reactive protein (CRP) (mg/dl). High-Sensitivity CRP was determined by immunonephelometry (mg/dl).
Change in Total fat mass (Kg), free fat mass (Kg) and visceral adipose tissue (Kg). | 0-30 days
  Body composition by dual-energy X-ray absorptiometry (DXA). Body composition was measured at baseline by DXA, using a Lunar Prodigy DEXA (GE Medical Systems, Waukesha, WI). Free Fat mass (Kg), Fat mass and visceral fat (Kg) data were derived from DXA using the DXA Prodigy enCORE software (version 17; GE Healthcare).
Change in inflammatory blood markers (ERS) (mm) | 0-30 days
  Inflammation markers in plasma: erythrocyte sedimentation rate (ESR) (mm). The erythrocyte sedimentation rate (ESR) was analyzed by capillary photometry (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, PhD, Principal Investigator — IRCCS Mondino Foundation, Pavia, 27100 Italy
Locations (1):
- Geriatric physical medicine and rehabilitation division at the Istituto Santa Margherita - Azienda di Servizi alla Persona di Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No